CLINICAL TRIAL: NCT02783898
Title: Randomised Controlled Trial of the Use of a Smart Phone Based Event Recorder Versus Standard Care for Patients Presenting to the Emergency Department With Palpitations and Pre-syncope
Brief Title: The IPED (Investigation of Palpitations in the ED) Study
Acronym: IPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/0153; R15/A164 (Other: Chest Heart Stroke Scotland); PG/17/63/33198 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2016-03-23; First posted 2016-05-26 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2018-03

CONDITIONS: Presyncope; Arrhythmias, Cardiac; Tachycardia, Supraventricular; Atrial Fibrillation
Keywords: pre syncope, palpitations
MeSH Terms: conditions — Syncope; Arrhythmias, Cardiac; Tachycardia, Supraventricular; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study (Experimental): All STUDY arm participants will be given an AliveCor Heart Monitor and trained in the use of the device. They will be followed up at 90 days. If a participants allocated to the Study arm, gets an episode of palpitations or pre-syncope and is able to record an AliveCor Heart Monitor ECG during the episode, the participant will email the ECG recorded by the AliveCor app directly to the study team. The study team will review the ECG. If specialist follow-up is not required the study team will inform the participant of this and ask them to arrange general practitioner follow up. If the participant records a serious significant arrhythmia during the study period, the study team will alert the participant immediately and refer them to the cardiac electrophysiology service.
  Interventions: Device: AliveCor Heart Monitor
- Control (No Intervention): All CONTROL arm participants will receive no other intervention. Participants in both groups will be admitted, referred or discharged by the treating clinician according to current hospital protocols. Participants in both groups will be followed up at 90 days through hospital electronic patient record (EPR) systems and through a standardised written questionnaire and follow-up telephone call including symptoms and contact with medical services, satisfaction and compliance.

INTERVENTIONS:
Device: AliveCor Heart Monitor — Smart phone based ECG event recorder
  Arms: Study

SUMMARY:
Palpitations (noticeable pounding, fluttering or irregular heart beat) and pre-syncope (near blackout) are common ED problems sometimes due to an abnormal cardiac rhythm. This is difficult to diagnose as examination and electrocardiogram (ECG) are commonly normal and symptoms have usually resolved by the time the patient arrives in the ED. Diagnosing an abnormal heart rhythm as the cause of symptoms rests on capturing it on an ECG and patients are usually discharged with advice to return to the ED again for a 12-lead ECG should symptoms recur. The investigators will recruit 242 adult participants to either study or control arms. All study arm participants will be given an AliveCor Heart Monitor and trained in the use of the device. Control arm participants will receive standard care only. Both groups will be followed-up at 90 days. The investigators believe a smart phone based event recorder will allow better and earlier diagnosis in patients with a compatible smart phone or tablet, and revolutionise ED care in this area.

DETAILED DESCRIPTION:
Palpitations (noticeable pounding, fluttering or irregular heart beat) and pre syncope (near blackout) are common ED problems sometimes due to an abnormal heart rhythm. Diagnosis is difficult as examination and electrocardiogram (ECG) are commonly normal and symptoms have usually resolved by the time the patient arrives in the ED. Diagnosing an abnormal heart rhythm as the cause of symptoms rests on capturing it on an ECG and patients are usually advised to return to the ED for a 12-lead ECG should symptoms recur. The investigators will recruit 242 participants aged 16 years or over presenting to the ED or Medical Assessment Unit of the Royal Infirmary of Edinburgh with an episode of palpitations or pre-syncope and who remain undiagnosed after ED assessment. The investigators will randomise and allocate participants to either study or control arms. All study arm participants will be given an AliveCor Heart Monitor and trained in the use of the device. Control arm participants will receive standard care only. If a participant allocated to the study arm has palpitations or pre-syncope during the 90-day study period, the participant can record an ECG using the AliveCor Monitor which can be viewed by the study team. Participants will be asked to log symptoms and whether the participant was able to record an ECG during the symptoms in a participant symptom diary, which the participant will return to the research team along with the Participant satisfaction and compliance questionnaire, and smart phone based event recorder at the end of the 90 days in a pre-paid stamped, addressed envelope. Participants will be phoned at 90 days to remind the participant to complete the Participant satisfaction and compliance questionnaire and to return this with the symptom diary and smart phone based event recorder. The investigators believe a smart phone based event recorder will allow better and earlier diagnosis in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participant aged 16 years or over
2. Participant presenting with an episode of palpitations or pre-syncope
3. Participant's underlying ECG rhythm during these episodes remains undiagnosed after clinical assessment.

Exclusion Criteria:

1. Prior diagnostic ECG
2. Palpitations or pre-syncope present during an admission ECG
3. Frequent episodes (i.e. at least once a day)
4. Participants under 16 years of age
5. Previous participation in the study
6. Inability or unwilling to give informed consent.
7. Participants with recent (i.e. within 3 months) myocardial infarction, severe heart failure (NYHA class 4) or unstable angina
8. Participants unwilling or unable to use the AliveCor Heart Monitor and AliveECG app
9. Participants without a compatible smart phone or tablet
10. Participants with cardiac pacemakers or other implanted electronic devices
11. No telephone number for follow-up
12. Participant in custody

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Reed, MA FRCEM MD, Principal Investigator — NHS Lothian
Locations (10):
- United Kingdom (10):
  - Royal Infirmary of Edinburgh, Edinburgh, Midlothian
  - Chesterfield, Chesterfield
  - Royal Devon and Exeter Hospital, Exeter
  - Leicester Royal Infirmary, Leicester
  - Royal London Hospital, Barts NHS Trust, London
  - Whipps Cross Hospital, Barts NHS Trust, London
  - Nottingham University Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Royal Berkshire Hospital, Reading
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiruganasambandamoorthy V, Taljaard M, Stiell IG, Sivilotti ML, Murray H, Vaidyanathan A, Rowe BH, Calder LA, Lang E, McRae A, Sheldon R, Wells GA. Emergency department management of syncope: need for standardization and improved risk stratification. Intern Emerg Med. 2015 Aug;10(5):619-27. doi: 10.1007/s11739-015-1237-1. Epub 2015 Apr 28. PMID 25918108
- [Background] Probst MA, Mower WR, Kanzaria HK, Hoffman JR, Buch EF, Sun BC. Analysis of emergency department visits for palpitations (from the National Hospital Ambulatory Medical Care Survey). Am J Cardiol. 2014 May 15;113(10):1685-90. doi: 10.1016/j.amjcard.2014.02.020. Epub 2014 Mar 1. PMID 24698469
- [Background] Lau JK, Lowres N, Neubeck L, Brieger DB, Sy RW, Galloway CD, Albert DE, Freedman SB. iPhone ECG application for community screening to detect silent atrial fibrillation: a novel technology to prevent stroke. Int J Cardiol. 2013 Apr 30;165(1):193-4. doi: 10.1016/j.ijcard.2013.01.220. Epub 2013 Mar 7. No abstract available. PMID 23465249
- [Background] Lowres N, Neubeck L, Salkeld G, Krass I, McLachlan AJ, Redfern J, Bennett AA, Briffa T, Bauman A, Martinez C, Wallenhorst C, Lau JK, Brieger DB, Sy RW, Freedman SB. Feasibility and cost-effectiveness of stroke prevention through community screening for atrial fibrillation using iPhone ECG in pharmacies. The SEARCH-AF study. Thromb Haemost. 2014 Jun;111(6):1167-76. doi: 10.1160/TH14-03-0231. Epub 2014 Apr 1. PMID 24687081
- [Background] Haberman ZC, Jahn RT, Bose R, Tun H, Shinbane JS, Doshi RN, Chang PM, Saxon LA. Wireless Smartphone ECG Enables Large-Scale Screening in Diverse Populations. J Cardiovasc Electrophysiol. 2015 May;26(5):520-6. doi: 10.1111/jce.12634. Epub 2015 Mar 19. PMID 25651872
- [Background] Tarakji KG, Wazni OM, Callahan T, Kanj M, Hakim AH, Wolski K, Wilkoff BL, Saliba W, Lindsay BD. Using a novel wireless system for monitoring patients after the atrial fibrillation ablation procedure: the iTransmit study. Heart Rhythm. 2015 Mar;12(3):554-559. doi: 10.1016/j.hrthm.2014.11.015. Epub 2014 Nov 18. PMID 25460854
- [Derived] Reed MJ, Grubb NR, Lang CC, O'Brien R, Simpson K, Padarenga M, Grant A, Tuck S, Keating L, Coffey F, Jones L, Harris T, Lloyd G, Gagg J, Smith JE, Coats T. Multi-centre Randomised Controlled Trial of a Smartphone-based Event Recorder Alongside Standard Care Versus Standard Care for Patients Presenting to the Emergency Department with Palpitations and Pre-syncope: The IPED (Investigation of Palpitations in the ED) study. EClinicalMedicine. 2019 Mar 3;8:37-46. doi: 10.1016/j.eclinm.2019.02.005. eCollection 2019 Feb. PMID 31193636
- [Derived] Reed MJ, Grubb NR, Lang CC, O'Brien R, Simpson K, Padarenga M, Grant A, Tuck S. Multi-centre randomised controlled trial of a smart phone-based event recorder alongside standard care versus standard care for patients presenting to the Emergency Department with palpitations and pre-syncope - the IPED (Investigation of Palpitations in the ED) study: study protocol for a randomised controlled trial. Trials. 2018 Dec 29;19(1):711. doi: 10.1186/s13063-018-3098-1. PMID 30594256

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 243 patients randomised. 1 participant removed after randomisation as did not meet inclusion criteria. 242 patients allocated to arms.
Period: Overall Study
Arm/Group | Study | Control
Started | 125 | 117
Completed | 124 | 116
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 125 | 117 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (14) | 39.1 (13.5) | 39.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 63 | 137
  Male | 51 | 54 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of presenting episode = Palpitations [Count of Participants; unit: Participants] | 110 | 109 | 219

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Rhythm Detection up to 90 Days
Description: Symptomatic rhythm detection rate of a smart phone based event recorder for symptomatic rhythm detection versus standard care.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
Participants | 69 | 11

2. Secondary Outcome: Number of Participants With Symptomatic Cardiac Rhythm Detection up to 90 Days
Description: Symptomatic rhythm detection rate of a smart phone based event recorder for cardiac arrhythmia detection versus standard care
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
Participants | 11 | 1

3. Secondary Outcome: Time to Detection of Symptomatic Rhythm
Description: Time to detection of symptomatic rhythm using a smart phone based event recorder versus standard care
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
days | 9.5 (16.1) | 42.9 (16)

4. Secondary Outcome: Time to Detection of Cardiac Arrhythmia Rhythm
Description: Time to detection of cardiac arrhythmia rhythm using a smart phone based event recorder versus standard care
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
days | 9.9 (15.6) | 48 (0)

5. Secondary Outcome: Number of Participants Treated or (Planned for Treatment) for Cardiac Arrhythmia
Description: Number of participants treated or (planned for treatment) for cardiac arrhythmia in participants using a smart phone based event recorder versus standard care
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
Participants | 12 | 6

6. Secondary Outcome: Number of Participants Finding the AliveCor Heart Monitor Easy to Use
Description: Number of Participants answering the participant questionnaire and finding the AliveCor heart monitor easy to use
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Study Group: The AliveCor heart monitor was easy to use
Arm/Group | Study Group
Number analyzed (Participants) | 125
Participants
  Strongly Agree | 48
  Agree | 32
  Missing | 33
  Strongly Disagree | 4
  Neutral | 8

7. Secondary Outcome: Financial Cost Per Diagnosis of Symptomatic Rhythm
Description: Financial cost per diagnosis of symptomatic rhythm using smart phone based event recorder versus standard care.
Time Frame: 90 days
Measure: Median (Full Range); unit: British pounds
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
British pounds | 474 [99 to 2697] | 1395 [0 to 4161]

8. Secondary Outcome: Number of Participants With Serious Outcome up to 90 Days
Description: Number of patients with all cause death and/or major adverse cardiac events (MACE; myocardial infarction, life threatening arrhythmia, insertion of pacemaker or internal cardiac defibrillator, insertion of pacing wire).
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study | Control
Number analyzed (Participants) | 124 | 116
Participants | 11 | 2

9. Secondary Outcome: Number of Participants Completing Questionnaire
Description: Measure of questionnaire compliance - Number of participants completing questionnaire
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Study Group: Questionnaire compliance
Arm/Group | Study Group
Number analyzed (Participants) | 125
Participants
  Completed questionnaire | 92
  Not completed | 33

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 0/124 | 1/116
Serious Adverse Events (participants affected / at risk) | 11/124 | 1/116
Other Adverse Events (participants affected / at risk) | 0/124 | 0/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study (N=124) | Control (N=116)
Major Adverse Cardiac Events (Cardiac disorders) | 11 (11) | 1 (1) — Number of patients with major adverse cardiac events (MACE; myocardial infarction, life threatening arrhythmia, insertion of pacemaker or internal cardiac defibrillator, insertion of pacing wire).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02783898/SAP_000.pdf
  • Study Protocol (2016-10-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT02783898/Prot_001.pdf